CLINICAL TRIAL: NCT01095835
Title: A Multicenter, Randomized, Controlled Study Comparing the Efficacy and Safety of 48 Weeks of 40kD Branched Pegylated Interferon Alfa-2a (PEG-IFN, RO 25-8310) Versus 96 Weeks of PEG-IFN, Alone or in Combination With 100 mg Lamivudine for 48 Weeks in Patients With HBeAg-Negative Chronic Hepatitis B
Brief Title: A Study of Pegylated Interferon Alfa-2a and Lamivudine in Patients With HBeAg-Negative Chronic Hepatitis B Virus (HBV)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML18253
Record Dates: First submitted 2010-03-26; First posted 2010-03-30 (Estimated); Results first posted 2016-11-03 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-03

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a; Lamivudine

ARMS (3):
- PEG-IFN48 (Experimental): Treatment with PEG-IFN in participants with HBeAg-negative chronic hepatitis B virus for 48 weeks.
  Interventions: Drug: Pegylated interferon (PEG-IFN) alfa-2a, 180 mcg
- PEG-IFN96 (Experimental): Treatment with PEG-IFN in participants with HBeAg-negative chronic hepatitis B virus for 48 weeks followed by another 48 weeks of PEG-IFN treatment (total 96 weeks of treatment).
  Interventions: Drug: Pegylated interferon (PEG-IFN) alfa-2a, 180 mcg; Drug: Pegylated interferon (PEG-IFN) alfa-2a, 135 mcg
- PEG-IFN+LAM96 (Experimental): Treatment with PEG-IFN and lamivudine in participants with HBeAg-negative chronic hepatitis B virus for 48 weeks followed by 48 weeks of only PEG-IFN treatment (total 96 weeks of treatment).
  Interventions: Drug: Pegylated interferon (PEG-IFN) alfa-2a, 180 mcg; Drug: Pegylated interferon (PEG-IFN) alfa-2a, 135 mcg; Drug: Lamivudine (LAM)

INTERVENTIONS:
Drug: Pegylated interferon (PEG-IFN) alfa-2a, 180 mcg — PEG-IFN alfa-2a 180 micrograms (mcg) was administered subcutaneously, once weekly from Week 0 to 48.
  Other Names: Pegasys®
Drug: Pegylated interferon (PEG-IFN) alfa-2a, 135 mcg — PEG-IFN alfa-2a 135 mcg was administered subcutaneously, once weekly from Week 49 to 96.
  Other Names: Pegasys®
  Arms: PEG-IFN+LAM96; PEG-IFN96
Drug: Lamivudine (LAM) — Lamivudine 100 milligrams (mg) was administered orally, daily from Week 0 to 48.
  Arms: PEG-IFN+LAM96

SUMMARY:
This study will compare the efficacy and safety of 2 different durations of treatment with pegylated interferon (PEG-IFN) alfa-2a in participants with Hepatitis B e Antigen (HBeAg)-negative chronic hepatitis B virus (HBV). It will also compare PEG-IFN alfa 2a treatment alone and in combination with lamivudine (LAM). The anticipated time on study treatment is 1-2 years, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adults 18-70 years of age;
* HBeAg-negative chronic hepatitis B for >/=6 months;
* liver disease consistent with chronic hepatitis B.

Exclusion Criteria:

* interferon-based, systemic anti-HBV, antiviral, anti-neoplastic, or immunomodulatory therapy </=12 months before first dose of study drug;
* non-responders to previous interferon therapy;
* co-infection with hepatitis A, C or D, or with human immunodeficiency virus (HIV);
* hepatocellular cancer;
* compensated (Child A, score 6) or decompensated liver disease (Child B or C).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2005-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- Italy (19):
  - Bari, Apulia
  - Castellana Grotte, Apulia
  - San Giovanni Rotondo, Apulia
  - Caserta, Campania
  - Napoli, Campania
  - Bologna, Emilia-Romagna
  - Parma, Emilia-Romagna
  - Reggio Emilia, Emilia-Romagna
  - Trieste, Friuli Venezia Giulia
  - Udine, Friuli Venezia Giulia
  - Brescia, Lombardy
  - Milan, Lombardy
  - Turin, Piedmont
  - Cagliari, Sardinia
  - Messina, Sicily
  - Palermo, Sicily
  - Pisa, Tuscany
  - Padua, Veneto
  - Verona, Veneto

REFERENCES:
- [Derived] Lampertico P, Vigano M, Di Costanzo GG, Sagnelli E, Fasano M, Di Marco V, Boninsegna S, Farci P, Fargion S, Giuberti T, Iannacone C, Regep L, Massetto B, Facchetti F, Colombo M; PegBeLiver Study Group. Randomised study comparing 48 and 96 weeks peginterferon alpha-2a therapy in genotype D HBeAg-negative chronic hepatitis B. Gut. 2013 Feb;62(2):290-8. doi: 10.1136/gutjnl-2011-301430. Epub 2012 Aug 2. PMID 22859496

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The Intent-to-Treat (ITT) population (n=128) included all participants randomized who received at least one dose of study medication. Three enrolled participants (total enrolled n=131) did not receive any study medication and were therefore excluded from the ITT population.The ITT population is reported in the Participant Flow.
Groups:
- PEG-IFN48: Treatment with pegylated interferon (PEG-IFN) alfa-2a in participants with HBeAg-negative chronic hepatitis B virus for 48 weeks. PEG-IFN alfa-2a 180 micrograms (mcg) was administered subcutaneously, once weekly from Week 0 to 48.
- PEG-IFN96: Treatment with PEG-IFN alfa-2a in participants with HBeAg-negative chronic hepatitis B virus for 48 weeks followed by another 48 weeks of PEG-IFN alfa-2a treatment (total 96 weeks of treatment). PEG-IFN alfa-2a 180 mcg was administered subcutaneously, once weekly from Week 0 to 48 followed by 135 mcg of PEG-IFN alfa-2a subcutaneously, once weekly from Week 49 to 96.
- PEG-IFN+LAM96: Treatment with PEG-IFN alfa-2a and lamivudine in participants with HBeAg-negative chronic hepatitis B virus for 48 weeks followed by 48 weeks of only PEG-IFN alfa-2a treatment (total 96 weeks of treatment). PEG-IFN alfa-2a 180 mcg subcutaneously, once weekly and 100 milligrams (mg) of oral lamivudine daily were administered from Week 0 to 48 followed by 135 mcg of only PEG-IFN alfa-2a, subcutaneously, once weekly from Week 49 to 96.
Period: Overall Study
Arm/Group | PEG-IFN48 | PEG-IFN96 | PEG-IFN+LAM96
Started | 51 | 52 | 25
Completed | 41 | 40 | 17
Not Completed | 10 | 12 | 8
Not completed — Adverse Event | 8 | 6 | 6
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 3 | 0
Not completed — Non study compliance | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Population: The ITT population included all participants randomized who received at least one dose of study medication.
Groups:
- PEG-IFN48: Treatment with PEG-IFN alfa-2a in participants with HBeAg-negative chronic hepatitis B virus for 48 weeks. PEG-IFN alfa-2a 180 micrograms (mcg) was administered subcutaneously, once weekly from Week 0 to 48.
- PEG-IFN+LAM96: Treatment with PEG-IFN alfa-2a and lamivudine in participants with HBeAg-negative chronic hepatitis B virus for 48 weeks followed by 48 weeks of only PEG-IFN alfa-2a treatment (total 96 weeks of treatment). PEG-IFN alfa-2a 180 mcg subcutaneously, once weekly and 100 mg of oral lamivudine daily were administered from Week 0 to 48 followed by 135 mcg of only PEG-IFN alfa-2a, subcutaneously, once weekly from Week 49 to 96.
- Total: Total of all reporting groups
Arm/Group | PEG-IFN48 | PEG-IFN96 | PEG-IFN+LAM96 | Total
Number analyzed (Participants) | 51 | 52 | 25 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (10.2) | 44.1 (10.4) | 45.6 (8.6) | 44.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 7 | 7 | 32
  Male | 33 | 45 | 18 | 96

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving the Combined Response at the End of the Follow-up Period
Description: Combined response was defined as alanine aminotransferase (ALT) normalization plus lowering of hepatitis B virus (HBV) deoxyribo nucleic acid (DNA) levels to <20,000 copies/mL (<3,400 IU/mL) and was measured at the end of the 48-week follow-up period. Participants with missing 48 weeks follow-up measurements were considered as non-responders. However, if the scheduled 48-weeks post-treatment tests were performed earlier or later than 48 weeks post-treatment, but not earlier than 36 weeks post-treatment, the corresponding results were considered to determine response.
Time Frame: At the end of the 48-week follow-up period at Week 144
Population: The ITT population included all participants randomized who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN48 | PEG-IFN96 | PEG-IFN+LAM96
Number analyzed (Participants) | 51 | 52 | 25
percentage of participants | 11.8 | 25.0 | 20.0
Statistical Analysis 1: Comparison: PEG-IFN48 vs PEG-IFN96; Test type: Superiority or Other; p = 0.08, Chi-squared

2. Secondary Outcome: Percentage of Participants Achieving the Combined Response at the End of Treatment
Description: Combined response was defined as ALT normalization plus lowering of HBV-DNA levels to <20,000 copies/mL (<3,400 IU/mL). In case of missing end of treatment measurements, the next available post-treatment value was used.
Time Frame: At end of treatment at Week 48 or 96 depending on the study arm
Population: The ITT population included all participants randomized who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN48 | PEG-IFN96 | PEG-IFN+LAM96
Number analyzed (Participants) | 51 | 52 | 25
percentage of participants | 29.4 | 38.5 | 32.0

3. Secondary Outcome: Percentage of Participants Achieving the Combined Response at 24 Weeks of Follow-up
Description: Combined response was defined as ALT normalization plus lowering of HBV-DNA levels to <20,000 copies/mL (<3,400 IU/mL). In case of missing week-24 post-treatment measurements, the nearest value with respect to the schedule time point in the time window 12 weeks post treatment until study end was used.
Time Frame: At the end of 24 weeks of follow-up at Week 120
Population: The ITT population included all participants randomized who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN48 | PEG-IFN96 | PEG-IFN+LAM96
Number analyzed (Participants) | 51 | 52 | 25
percentage of participants | 23.5 | 28.8 | 24.0

4. Secondary Outcome: Percentage of Participants Achieving Combined Response Using a Cut-Off for HBV-DNA Levels to 2,000 IU/mL
Description: Combined response was defined here as ALT normalization plus lowering HBV-DNA levels to a cutt-off <2,000 IU/mL. In case of missing end of treatment measurements, the next available post-treatment value was used. In case of missing week-24 post-treatment measurements, the nearest value with respect to the schedule time point in the time window 12 weeks post treatment until study end was used. Participants with missing 48 weeks follow-up measurements were considered as non-responders. However, if the scheduled 48-weeks post-treatment tests were performed earlier or later than 48 weeks post-treatment, but not earlier than 36 weeks post-treatment, the corresponding results were considered to determine response.
Time Frame: At end of treatment at Week 48 or 96 depending on the study arm, at the end of 24 weeks of follow-up at Week 120 and at the end of the follow-up period at Week 144
Population: The ITT population included all participants randomized who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN48 | PEG-IFN96 | PEG-IFN+LAM96
Number analyzed (Participants) | 51 | 52 | 25
percentage of participants
  End of treatment | 29.4 | 38.5 | 28.0
  24 weeks of follow-up | 21.6 | 26.9 | 20.0
  48 weeks of follow-up | 11.8 | 23.1 | 20.0

5. Secondary Outcome: Percentage of Participants Achieving Histological Response
Description: Histological response was defined as an improvement by >/= 2 in the Necroinflammatory Grading and/or by an improvement by >/= 1 score in Fibrosis Staging according to Ishak. Necroinflammatory Grading ranges 0-14 and is the combined score for necrosis, range 0-10 and inflammation, range 0-4. The participant is scored for only one inflammatory condition. A higher score indicates worse condition. Fibrosis Staging according to Ishak ranges 0-6 and a higher score indicates greater fibrosis.
Time Frame: At the end of the 48-week follow-up period at Week 144
Population: The ITT population included all participants randomized who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN48 | PEG-IFN96 | PEG-IFN+LAM96
Number analyzed (Participants) | 51 | 52 | 25
percentage of participants | 13.7 | 5.8 | 8.0

6. Secondary Outcome: Change From Baseline of Quantitative Hepatitis B Surface Antigen (HbsAg) Level at the End of Treatment
Time Frame: At the end of treatment at Week 48 or 96 depending on the study arm
Population: The ITT population included all participants randomized who received at least one dose of study medication. Baseline values are included for those participants for whom a baseline value was measured. Change from baseline values includes only those participants with both a baseline value and a value for the summarized time period.
Measure: Mean (Standard Deviation); unit: IU/mL
Arm/Group | PEG-IFN48 | PEG-IFN96 | PEG-IFN+LAM96
Number analyzed (Participants) | 51 | 52 | 25
IU/mL
  Baseline (n=51, 51, 25) | 9642.6 (19756.4) | 7229.8 (6459.0) | 8981.0 (7728.5)
  Change from baseline (n=44, 44, 20) | -2801.1 (14691.2) | -2282.1 (6007.1) | -3121.2 (7128.9)

7. Secondary Outcome: Percentage of Participants With Lamivudine Genotype Resistance During PEG-IFN+LAM96 Combined Therapy
Description: Lamivudine resistance mutations were assessed by detection of the following mutations: rtL80V, rtL80I, rtV173G, rtV173L, rtL180M, rtA181T, rtA181V, rtM204V, rtM204I and rtN236T.
Time Frame: At the end of the treatment period at Week 96
Population: The ITT population for arm PEG-IFN+LAM96 included all participants randomized to PEG-IFN+LAM96 who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN+LAM96
Number analyzed (Participants) | 25
percentage of participants | 0

8. Other Pre Specified Outcome: Percentage of Participants With ALT Normalization
Time Frame: as for outcome 4
Population: The ITT population included all participants randomized who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN48 | PEG-IFN96 | PEG-IFN+LAM96
Number analyzed (Participants) | 51 | 52 | 25
percentage of participants
  End of treatment | 35.3 | 40.4 | 40.0
  24 weeks of follow-up | 45.1 | 46.2 | 40.0
  48 weeks of follow-up | 35.3 | 34.6 | 36.0

9. Other Pre Specified Outcome: Percentage of Participants With HBV-DNA Lowering to <3,400 IU/mL and to < 2,000 IU/mL
Time Frame: as for outcome 4
Population: The ITT population included all participants randomized who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN48 | PEG-IFN96 | PEG-IFN+LAM96
Number analyzed (Participants) | 51 | 52 | 25
percentage of participants
  End of treatment: HBV-DNA < 3,400 IU/mL | 60.8 | 67.3 | 76.0
  24 weeks of follow-up: HBV-DNA < 3,400 IU/mL | 23.5 | 30.8 | 24.0
  48 weeks of follow-up: HBV-DNA < 3,400 IU/mL | 11.8 | 30.8 | 20.0
  End of treatment: HBV-DNA < 2,000 IU/mL | 58.8 | 67.3 | 72.0
  24 weeks of follow-up: HBV-DNA < 2,000 IU/mL | 21.6 | 28.8 | 20.0
  48 weeks of follow-up: HBV-DNA < 2,000 IU/mL | 11.8 | 28.8 | 20.0

10. Other Pre Specified Outcome: Percentage of Participants With HBV-DNA Below Limit of Quantification
Description: HBV-DNA limit < 6 IU/mL was defined as below quantification.
Time Frame: as for outcome 4
Population: The ITT population included all participants randomized who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN48 | PEG-IFN96 | PEG-IFN+LAM96
Number analyzed (Participants) | 51 | 52 | 25
percentage of participants
  End of treatment | 17.6 | 30.8 | 24.0
  24 weeks of follow-up | 0.0 | 7.7 | 4.0
  48 weeks of follow-up | 2.0 | 7.7 | 8.0

11. Other Pre Specified Outcome: Percentage of Participants With Loss of Hepatitis B Surface Antigen (HbsAg) and Hepatitis B Surface Antibodies (Anti-HBs) Seroconversion
Description: This outcome measure presents percentage of participants with a combined response of HBsAg < 5 IU/mL and anti-HBs positive. Positive anti-HBs represents antibodies produced against Hepatitis B Surface Antigen (HBsAg) and is an indication of recovery and immunity from HBV infection.
Time Frame: as for outcome 4
Population: The ITT population included all participants randomized who received at least one dose of study medication.
Measure: Number; unit: percentage of participants
Arm/Group | PEG-IFN48 | PEG-IFN96 | PEG-IFN+LAM96
Number analyzed (Participants) | 51 | 52 | 25
percentage of participants
  End of treatment | 2.0 | 3.8 | 0.0
  24 weeks of follow-up | 0.0 | 5.8 | 0.0
  48 weeks of follow-up | 0.0 | 7.7 | 0.0

ADVERSE EVENTS:
Time Frame: Up to 48 weeks after last study treatment dose (up to Week 144)
Description: The Safety population included all participants randomized who received at least one dose of study medication and had at least one post-baseline safety assessment. In addition to participants excluded from the Intent-to-Treat (ITT) population, one participant in the ITT population did not perform a post-baseline safety assessment, and was therefore excluded from the safety population.
Groups:
- PEG-IFN + LAM96: Treatment with PEG-IFN alfa-2a and lamivudine in participants with HBeAg-negative chronic hepatitis B virus for 48 weeks followed by 48 weeks of only PEG-IFN alfa-2a treatment (total 96 weeks of treatment). PEG-IFN alfa-2a 180 mcg subcutaneously, once weekly and 100 milligrams (mg) of oral lamivudine daily were administered from Week 0 to 48 followed by 135 mcg of only PEG-IFN alfa-2a, subcutaneously, once weekly from Week 49 to 96.
Arm/Group | PEG-IFN48 | PEG-IFN96 | PEG-IFN + LAM96
Serious Adverse Events (participants affected / at risk) | 7/50 | 3/52 | 6/25
Other Adverse Events (participants affected / at risk) | 25/50 | 27/52 | 13/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN48 (N=50) | PEG-IFN96 (N=52) | PEG-IFN + LAM96 (N=25)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 0
Infected cyst (Infections and infestations) | 0 | 0 | 1
Facial palsy (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PEG-IFN48 (N=50) | PEG-IFN96 (N=52) | PEG-IFN + LAM96 (N=25)
Anaemia (Blood and lymphatic system disorders) | 5 | 4 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 3 | 0
Neutropenia (Blood and lymphatic system disorders) | 12 | 9 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 6 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 4 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 3 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 4 | 2
Nausea (Gastrointestinal disorders) | 5 | 2 | 2
Asthenia (General disorders) | 17 | 19 | 11
Influenza like illness (General disorders) | 9 | 10 | 4
Pyrexia (General disorders) | 18 | 19 | 8
Pharyngitis (Infections and infestations) | 3 | 2 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 2
Urinary tract infection (Infections and infestations) | 3 | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 4 | 2
Blood thyroid stimulating hormone increased (Investigations) | 1 | 0 | 2
Platelet count decreased (Investigations) | 0 | 4 | 0
White blood cell count decreased (Investigations) | 0 | 3 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 6 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 6 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 6 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 8 | 4
Headache (Nervous system disorders) | 13 | 8 | 7
Sciatica (Nervous system disorders) | 1 | 3 | 0
Anxiety (Psychiatric disorders) | 4 | 5 | 2
Insomnia (Psychiatric disorders) | 4 | 0 | 2
Irritability (Psychiatric disorders) | 0 | 3 | 2
Nervousness (Psychiatric disorders) | 0 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 6 | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 2
Hypertension (Vascular disorders) | 1 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.